CLINICAL TRIAL: NCT03836534
Title: Multicentric Prospective Study of the Observance of Outpatient Treatments in Reims During the Care Continuum
Brief Title: the Observance of Emergency Exit Treatments During the Stay of Care at the Exit of Reims Emergencies
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18168
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Patient Coming to the Emergency Department for Any Reason

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient coming to the emergency department: the group studied only concern adult adults consulting in the emergency departments and leaving after their consultations, during the permanence of care
  Interventions: Behavioral: adherence to treatment of patients coming out of emergencies

INTERVENTIONS:
Behavioral: adherence to treatment of patients coming out of emergencies — Phone contact of patients within 48 hours of the consultation

SUMMARY:
The investigators would like to include patients consulting in a Accident and Emergency Department (AED) during the permanence of care the week of March 11 to 17, 2018. The data collection would concern socio-demographic data, their consultation to the AED, the follow-up given to the consultation and would take place by telephone contact of patients within 48 hours of the consultation.

why patients come to the emergency room, what are they waiting for? what are their main motivations? what do they do in emergencies, do they follow the treatments and recommendations?

DETAILED DESCRIPTION:
Study of the observance of emergency exit treatments during the permanence of care. This is a descriptive study with a prospective data collection that does not alter the management of the patient. The study is epidemiological, cross-sectional, prospective inclusion.

The investigators would like to include patients consulting in a AED during the permanence of care the week of March 11 to 17, 2018. The data collection would concern socio-demographic data, their consultation to the AED, the follow-up given to the consultation and would take place by telephone contact of patients within 48 hours of the consultation.

The objective is to study the follow-up given by the consultation to the emergencies, in terms of compliance, follow-up of the recommendations, the objective sought by the patient coming to the emergency department.

Understand the motivation of the consultation and why the treatment was not followed where appropriate.

Is there a sociodemographic explanation or is it the health network that results in the saturation of emergency services? Does the system still meet the expectations of people using it?

ELIGIBILITY:
Inclusion Criteria:

* adults
* consultation during the early stages of care
* leaving after consultation
* agrees to participate in the study

Exclusion Criteria:

* minor patients
* permanently off care
* hospitalized patients
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the group studied only concern adults consulting in the emergency and leaving after their consultations, durning the permanence of care
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
adherence to treatment | 2 days
  Number of Participants who visited of the drugstore after emergency visit

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided